CLINICAL TRIAL: NCT04140071
Title: NutriQuébec: a Unique Web-based Prospective Cohort Study to Monitor the Population's Eating Habits in the Province of Québec.
Brief Title: NutriQuébec: a Web-based Prospective Cohort Study to Monitor the Population's Eating Habits in the Province of Québec.
Status: Recruiting | Type: Observational
Sponsor: Laval University (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-042 Phase II A3/ 14-05-20
Record Dates: First submitted 2019-10-07; First posted 2019-10-25 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Eating Habits
Keywords: Eating habits; Web-based prospective cohort study; Lifestyle habits; Health; Diet quality
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The epidemic of non-communicable diseases such as cardiovascular diseases and type 2 diabetes is attributable in large part to unhealthy eating habits and physical inactivity. In the Fall of 2016, the Québec Government launched its first-ever Government Health Prevention Policy (PGPS) to act on a set of factors to improve the health status and quality of life of the population of Quebec and to reduce social inequalities in health. NutriQuébec is a web-based prospective cohort study whose primary aim is to quantify the impact of the implementation of the PGPS on the Québec population's eating habits over the years.

NutriQuébec will recruit over the next 3 years 20,000 adults living in the Province of Québec in Canada through a vast multimedia campaign designed to reach different segments of the population, including subgroups with a low socioeconomic status. Participants will be invited to complete on a web-based platform nine core questionnaires on a yearly basis. Questionnaires will assess several dimensions related to lifestyle, including eating habits and physical activity habits, as well as a large number of personal characteristics and global health status. The time course of the changes in eating habits will be analyzed in conjecture with the implementation of the PGPS to quantify its impact at a population level. Data will be analyzed while accounting for sociodemographic weight of participants, to achieve representativeness of the adult Québec population.

NutriQuébec will provide essential data for the long-term evaluation of eating habits after Québec's PGPS is launched.

DETAILED DESCRIPTION:
NutriQuébec is an open cohort with continuous and uninterrupted recruitment over the study duration, which is currently funded until 2022. The target sample size is 20,000 adults based on a non-probability sampling. A vast multimedia campaign will be deployed to reach the target population throughout the province of Québec. More specifically, television, radio and print interviews will be organized periodically. Key leading figures in the area of food and health will be solicited to promote the project on various media platforms. The project will also be publicized on social networks, including on the NutriQuébec Facebook page. The Québec Government and several of its community partners will be invited to promote NutriQuébec via their website, newsletters and/or the social networks they use. In addition, recruitment ads will be distributed through several channels, including: 1) email lists from partners and universities in Québec; and 2) public places such as community centers, health institutions and companies. All of the above-mentioned recruitment methods will invite individuals interested in the study to visit the NutriQuébec website for more information and to register.

After having created an account on the secured PULSAR platform, each individual will be invited to provide informed consent to participate in the project.Their eligibility (age and address of residence) will be automatically verified at registration. Once registered and having consented, participants will be invited through email to complete the core questionnaires by logging into their personal and secured account.

Core questionnaires will be completed on a yearly basis, based on the date of the participants' first registration. These core questionnaires assess lifestyle habits including eating habits, physical activity habits, sleep quality, tobacco, alcohol and drug habits as well as personal characteristics, food security and health status.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 and over with a residential address in Québec (Canada)
* Be able to read and understand French or English
* Have access to Internet (with a computer or an electronic tablet)
* Have an active email address

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults living in the province of Québec (Canada)
Sampling Method: Non-Probability Sample
Enrollment: 20000 (Estimated)
Dates: Start 2019-06-26 (Actual); Primary Completion 2043-06-25 (Estimated); Study Completion 2043-06-25 (Estimated)

PRIMARY OUTCOMES:
Vegetable and fruit intakes | Annual, ongoing assessment (up to 25 years of follow-up)
  Vegetable and fruit intakes will be assessed from the average of 3 validated Web-based 24-hour recalls. Vegetable and fruit intakes will be reported as the number of times consumed per day.

SECONDARY OUTCOMES:
Diet quality | Annual, ongoing assessment (up to 25 years of follow-up)
  Diet quality will be assessed from the average of 3 validated Web-based 24-hour recalls using the Canadian Health Eating Index on a scale of 0-100.

CONTACTS AND LOCATIONS:
Overall Officials: Benoît Lamarche, PhD, Principal Investigator — Laval University
Locations (1):
- Laval University, Québec, Canada

REFERENCES:
- [Derived] Rochette M, Rochefort G, Laramee C, Lapointe A, Lemieux S, Belanger-Gravel A, Desroches S, Provencher V, Lamarche B. Local food procurement behavior and overall diet quality among adults in Quebec: results from the NutriQuebec project. Nutr J. 2024 Nov 14;23(1):143. doi: 10.1186/s12937-024-01045-w. PMID 39543697
- [Derived] Lapointe A, Laramee C, Belanger-Gravel A, Buckeridge DL, Desroches S, Garriguet D, Gauvin L, Lemieux S, Plante C, Lamarche B. NutriQuebec: a unique web-based prospective cohort study to monitor the population's eating and other lifestyle behaviours in the province of Quebec. BMJ Open. 2020 Oct 28;10(10):e039889. doi: 10.1136/bmjopen-2020-039889. PMID 33115902